CLINICAL TRIAL: NCT04858009
Title: A Phase II Study of Hyperthermic Intraperitoneal Chemotherapy (HIPEC) for Patients With Pancreatic Cancer and Peritoneal Metastasis
Brief Title: Hyperthermic Intraperitoneal Chemotherapy for the Treatment of Pancreatic Cancer and Peritoneal Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cornelius A. Thiels, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-009451; NCI-2021-02990 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-04-14; First posted 2021-04-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Pancreatic Carcinoma; Stage IV Pancreatic Cancer AJCC v8; Metastatic Malignant Neoplasm in the Peritoneum
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Hyperthermic Intraperitoneal Chemotherapy; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (HIPEC) (Experimental): Patients undergo HIPEC with nab-paclitaxel and cisplatin over 90 minutes in the absence of disease progression or unacceptable toxicity. Patients may undergo additional HIPEC with paclitaxel and cisplatin up to 5 times. Patients undergo CT scan, MRI or PET during screening.
  Interventions: Drug: Cisplatin; Drug: Hyperthermic Intraperitoneal Chemotherapy; Drug: Nab-paclitaxel; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Cisplatin — Given via HIPEC
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Hyperthermic Intraperitoneal Chemotherapy — Undergo HIPEC with mitomycin and cisplatin
  Other Names: HIPEC
Drug: Nab-paclitaxel — Given via HIPEC
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Paclitaxel nanoparticle albumin-bound; Protein-bound Paclitaxel
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized Tomography; CT; CT Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; Nuclear magnetic resonance imaging (NMRI); Structural MRI (sMRI)
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; positron emission tomography scan; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial studies the effects of hyperthermic intraperitoneal chemotherapy (HIPEC) in treating patients with pancreatic cancer that has spread to the internal abdominal area (peritoneal metastasis). Chemotherapy drugs, such as nab-paclitaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. HIPEC involves "heated" chemotherapy that is placed directly in the abdomen through laparoscopic instruments, instead of through an intravenous injection. This study may help doctors determine how safe and effective HIPEC work in treating patient with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate overall survival and disease-free survival outcomes for patients with pancreatic adenocarcinoma with limited low volume peritoneal metastasis or positive peritoneal cytology undergoing hyperthermic intraperitoneal chemotherapy.

SECONDARY OBJECTIVE:

I. To assess morbidity for patients with pancreatic adenocarcinoma with limited low volume peritoneal metastasis or positive peritoneal cytology undergoing hyperthermic intraperitoneal chemotherapy.

OUTLINE:

Patients undergo HIPEC with nab-paclitaxel and cisplatin over 90 minutes in the absence of disease progression or unacceptable toxicity. Patients may undergo additional HIPEC with paclitaxel and cisplatin up to 5 times. Patients undergo computed tomography (CT) scan, magnetic resonance imaging (MRI) or positron emission tomography (PET) during screening.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 but =< 80
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Cytologic or histologic proof of adenocarcinoma of the pancreas
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 60,000/Ul
* Serum creatinine =< 1.5 mg/dL
* Distant metastatic disease of peritoneum may be visualized on imaging:

  * Positive peritoneal cytology
  * Limited carcinomatosis on diagnostic laparoscopy or laparotomy
  * KRASD assay positive peritoneal washings/cytology
* Completion of preoperative systemic chemotherapy with biochemical, metabolic, and/or radiographic response defined as a reduction in the baseline CA 19-9 by > 50% or radiographic response as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or metabolic response on positron emission tomography (PET)-magnetic resonance imaging (MRI) defined by PET Response Criteria in Solid Tumors (PERCIST) criteria
* Peritoneal Carcinomatosis Index (PCI) =< 7 and surgeons deems high likelihood for a complete cytoreduction

Exclusion Criteria:

* Distant metastatic disease not limited to peritoneum:

  * Solid organ metastases (liver, central nervous system, lung)
* Infections such as pneumonia or wound infections that would preclude protocol therapy
* Women with a positive urine or serum pregnancy test are excluded from this study; women of childbearing potential (defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to refrain from breast feeding and practice adequate contraception as specified in the informed consent. Adequate contraception consists of oral contraceptive, implantable contraceptives, injectable contraceptives, a double barrier method, or abstinence
* Subjects deemed unable to comply with study and/or follow-up procedures
* Subjects with a known hypersensitivity to protocol systemic chemotherapy that was life-threatening, required hospitalization or prolongation of existing hospitalization, or resulted in persistent or significant disability or incapacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 4 years
  Overall survival will be assessed from the date of cytoreduction and hyperthermic intraperitoneal chemotherapy (HIPEC) to death by any cause, regardless of disease recurrence. Patterns of tumor recurrence and survival will be assessed by reviewing routine surveillance imaging. Patient may be contacted by telephone and/or videoconferencing.
Progression-free survival | Up to 4 years
  Progression-free survival is will be assessed from the date of cytoreduction and HIPEC to recurrence of tumor or death. Patterns of tumor recurrence and survival will be assessed by reviewing routine surveillance imaging. Patient may be contacted by telephone and/or videoconferencing.

SECONDARY OUTCOMES:
Morbidity | 30 days; up to 4 years
  Morbidity is the state of having a specific illness or condition. Morbidity will be measured based on hospital length of stay, readmission rate, reoperation rate, and 30-day mortality (death).

CONTACTS AND LOCATIONS:
Overall Officials: Cornelius A. Thiels, DO, MBA, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Gudmundsdottir H, Yonkus JA, Thiels CA, Warner SG, Cleary SP, Kendrick ML, Truty MJ, Grotz TE. Oncologic Outcomes of Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy for Highly Selected Patients with Metastatic Pancreatic Ductal Adenocarcinoma. Ann Surg Oncol. 2023 Nov;30(12):7833-7839. doi: 10.1245/s10434-023-14138-3. Epub 2023 Aug 19. PMID 37596449
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials